CLINICAL TRIAL: NCT00306436
Title: Evaluation of the Impact of a Comprehensive Clinical Management on the Quality of Blood Pressure and Glycemic Control in Diabetic Uremic Patients
Brief Title: Comprehensive Management of Diabetic Patients With Renal Impairment : Impact on Blood Pressure and Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 9286-01; 2001-027
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetes; renal deficiency; hypertension
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: comprehensive management

SUMMARY:
Diabetes is the leading cause of end-stage renal disease in developed countries. Hypertension and metabolic control are known to affect the progression of renal deficiency and patient's outcome. Our project aims at implementing a multidisciplinary and systematic approach of diabetic patients with renal deficiency, and at evaluating the impact of metabolic and blood pressure targets as recommended by current guidelines.

DETAILED DESCRIPTION:
Complications of diabetes are influenced by the quality of blood pressure control and of metabolic control. Several prospective studies have shown a positive effect of the implementation of such control, however metabolic and blood pressure targets are not achieved for about 30% of diabetic uremic patients.

Our project aims at evaluating a comprehensive management approach of diabetic patients affected by renal insufficiency, defined by glomerular filtration rate (GRF) <60 mL/min/1,73 m², through an alternate and complementary follow-up by the nephrologist and the diabetologist.

During a first period (one year), patients are managed as "usually". After this period, the patients will start the multidisciplinary health care during at least two years. They will be followed-up by the diabetologist every 4 months. According to his GFR measured by renal clearance of Cr-EDTA, the patient will be followed-up by the nephrologist every year if the GFR is between 60 and 40 ml/min, every 4 months if the GFR is between 40 and 20 ml/min, and every 1 or 2 months if the GFR is under 20 ml/min. GFR will be re-evaluated every year (Cr-EDTA or Cockcroft-Gault formula) and so medical examination frequency. Guidelines will be applied regarding blood pressure control (objective: < 135/85 mmHg, and < 125/75 mmHg if proteinuria > 1g/24H, choice of drugs, implementation of the treatment...) and glycemic control (current guidelines according to the French Health Technology Information Agency, ANAES). Another important component of the management will be the implementation of nutritional balance and foot care.

Every two years, a detailed nutritional checkup will be planned by the diabetologist and a cardiologic check-up will be planned by the nephrologist during one day in the local nephrology department.

A biobank will be built up after patient's consent. We will assess the impact of this intervention (guidelines application + multidisciplinary methodical and complementary follow-up) in terms of glycemic and blood pressure control.

The percentage of patients who will obtain a good glycemic and blood pressure control will be analysed and compared between the two follow-up period (before/after the intervention).

If validated this strategy may provide the basis of a care network focused on an optimum diabetic health care.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients affected by renal insufficiency defined by glomerular filtration rate < 60 ml/min/1,73 m² by the Cockcroft-Gault formula
* signed informed consent

Exclusion Criteria:

* pregnant woman
* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
composite criteria reflecting a good glycemic and arterial pressure status. Success defined by all measurements of HbA1c < 6.5% and of systolic (diastolic) pressure <=135 (85) mmHg if proteinuria is < 1g/24h or <= 125 (75) if proteinuria is => 1g/24h

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lasseur, Doctor, Principal Investigator — University Hospital, Bordeaux; Geneviève Chêne, Professor, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service de Néphrologie-Hémodialyse du Pr C.Combe, Hôpital Pellegrin, Place Amélie Raba-Léon, Bordeaux, France